CLINICAL TRIAL: NCT03734692
Title: Systemic Immune Checkpoint Blockade and Intraperitoneal Chemo-Immunotherapy in Recurrent Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert Edwards (Other)
Collaborators: AIM ImmunoTech Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Robert Edwards, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 18-087
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — poly(I).poly(c12,U); pembrolizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- cisplatin + rintatolimod + pembrolizumab (Experimental): Intraperitoneal (IP) cisplatin 50mg/m^2 solution with IP rintatolimod 200 mg solution and IV pembrolizumab 200 mg solution.
  Interventions: Drug: Rintatolimod; Drug: Pembrolizumab; Drug: Cisplatin

INTERVENTIONS:
Drug: Rintatolimod — 200 mg by IP administration over 1-2 hours
  Other Names: Ampligen
Drug: Pembrolizumab — 200 mg will be administered as a 30 minute IV infusion
  Other Names: Keytruda
Drug: Cisplatin — 50mg/m^2 solution
  Other Names: Platinol

SUMMARY:
This is a phase II single arm efficacy/safety trial that will evaluate the effectiveness of combining intensive locoregional intraperitoneal (IP) chemoimmunotherapy of cisplatin with IP rintatolimod (TLR-3 agonist) and IV infusion of the checkpoint inhibitor pembrolizumab (IVP) for patients with recurrent platinum-sensitive ovarian cancer (OC).

DETAILED DESCRIPTION:
Patients will receive a total of six treatment cycles, at 3-week intervals. The study will use an IP neoadjuvant approach (IP chemoimmunotherapy of cisplatin with IP rintatolimod and IV infusion of pembrolizumab), followed by interval cytoreduction (usually laparoscopically) of residual tumor. Cytoreduction will occur approximately 4 weeks after the fourth treatment cycle. Post-surgery the investigators will consolidate with 2 additional courses of same chemo-immunotherapy regimen. Catheter will be removed 12 weeks after the last treatment. All surgical procedures, if done laparoscopically, are outpatient and will yield up to three serial biopsies of the tumor sites: 1) at catheter placement; 2) at interval cytoreduction which consists of removal of any visible tumor sites and the site biopsied initially whether tumor is present or not; 3) at catheter removal, when site of first tumor biopsy will be re-biopsied for pathologic response.

ELIGIBILITY:
Inclusion Criteria :

1. Patients must be at least 18 years of age on the day of signing informed consent.
2. Patients must have first or second peritoneal recurrence of epithelial adenocarcinoma or carcinosarcoma of ovarian, tubal or peritoneal origin:

   1. Histologic documentation of the original primary tumor is required via the pathology report.
   2. Original tumor blocks from the primary diagnosis will be requested by our study pathologist at Magee-Women's Hospital of UPMC Cancer Centers if the patient did not have their initial surgery at Magee. Original tumor blocks may be reviewed after registration (informed consent and enrollment). Tumor block should be held until study is completed.
3. Patients must have completed prior platinum-based therapy. Response can be complete or partial if it otherwise meets platinum sensitive criteria, see below.
4. Patients must be platinum-sensitive, defined as having a progression free interval (PFI) of more than 6 months (180 days) from any platinum therapy. Patients are allowed to have had other lines of therapy since last platinum if PFI after platinum therapy meets platinum sensitive criteria.
5. Patients must have measurable disease in the peritoneal cavity, measurable per RECIST 1.1 criteria:

   1. A mass with a length of 1.0 cm or greater and/or
   2. A lymph node with a length of 1.5 cm or greater in the shortest axis.
6. Patients must be a reasonable candidate for laparoscopy and IP platinum regimen with no prior evidence of clinically significant intra-abdominal adhesions, persistent abdominal wall infections, renal toxicity or bowel obstruction.
7. Patients of childbearing potential must:

   1. Have a negative pregnancy test prior to the study entry.
   2. Must discontinue breastfeeding prior to the first date of treatment on this study if applicable.
   3. Agree to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
8. Patients must agree to the protocol designated clinical monitoring to receive the study regimens.
9. The participant provides written informed consent for the trial.
10. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 28 days prior to the date of allocation/randomization.
11. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 28days prior to the start of study treatment.

Exclusion Criteria :

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to infusion of treatment regimen (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

   * Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
   * Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Patients with previous pelvic radiation therapy.
6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   o Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Patients with tumors of low malignant potential, except ovarian pseudomyxomas, or with no peritoneal disease.
10. Concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated basal or squamous cell carcinoma, non- melanomatous skin cancer or curatively resected cervical cancer or per physician discretion that the previous cancer was adequately treated with curative intent and unlikely to recur (the study PI must concur with this determination).
11. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
12. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
13. Has a known allergy to cisplatin chemotherapy. Patients with carboplatin allergy may be included if they tolerate a test dose of IV cisplatin given in monitored floor conditions.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
16. Has an active infection requiring systemic therapy.
17. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
18. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA qualitative is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
19. Has a known history of active TB (Bacillus Tuberculosis)
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Is pregnant or breastfeeding, or expecting to conceive or within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer is limited to the female population.
Enrollment: 24 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2027-01-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edwards, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 68.0 [51.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Disease.Site.Diagnosis [Count of Participants; unit: Participants]
  Malignant neoplasm of fallopian tube | 2
  Malignant neoplasm of ovary | 2
  Ovary | 20
Histology [Count of Participants; unit: Participants]
  ADENOCARCINOMA IN SITU, NOS | 1
  ADENOCARCINOMA, METASTATIC, NOS | 1
  ADENOCARCINOMA, NOS | 10
  CARCINOMA IN SITU, NOS | 2
  CARCINOMA, NOS | 4
  MULLERIAN MIXED TUMOR | 1
  PAPILLARY CARCINOMA, NOS | 1
  SEROUS ADENOCARCINOFIBROMA | 1
  Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The proportion of subjects with the best response of complete response (CR), or partial response (PR) per Response Evaluation Criteria for Solid Tumors (RECIST 1.1). Per RECIST 1.1 , CR is defined as all target lesions gone; PR is defined as a > 30% decrease in size of lesion from baseline.
Time Frame: At 13 weeks
Population: Treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 24
percentage of patients | 50 [31 to 69]

2. Secondary Outcome: DLTs Related to Treatment
Description: Number of patients who experience Adverse Events per CTCAE v5.0 related to study treatment, including any death not clearly due to disease or extraneous causes, AE leading to a dose delay of greater than 14 days in initiation of cycle 2, a DLT occurring during Cycle 1 of treatment: Grade ≥ 3 renal toxicity, diarrhea, skin toxicity, injection site reactions, anaphylaxis, hematologic toxicities lasting more than 48 hours (including neutropenia), non-hematologic toxicities, neurological symptoms, thrombocytopenia and hemorrhage, liver function test increase; Grade ≥ 2 or greater bronchospasm, allergic reaction or generalized urticaria, autoimmune reaction, pneumonitis; Fever > 41°C, uncontrolled for over 4 hours in the absence of a medical cause Evaluation of liver toxicity per Hy's Law: Drug causes hepatocellular injury (higher incidence of 3-fold or greater elevations above the ULN of ALT or AST); Total Bilirubin>2xULN (without initial cholestasis (elevated serum alkaline phosphatase)
Time Frame: At baseline (pre-treatment) and at 12 weeks (after the start of treatment)
Population: Treated patients monitored for DLTs.
Measure: Number; unit: patients
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 24
patients | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: The length of time during and after study treatment that a patient does not experience worsening disease. Per RECIST 1.1 or dies from any cause. Progression is defined as a > 20% increase from smallest sum of longest (lesion) diameter recorded since treatment started (best response - target lesions) and/or, enlargement of non-target lesions.
Time Frame: up to 4 years
Reporting Status: Not Posted

4. Secondary Outcome: Time To Disease Progression
Description: The length of time during and after study treatment that a patient remains alive without worsening disease. Per RECIST 1.1, progression is defined as a > 20% increase from smallest sum of longest (lesion) diameter recorded since treatment started (best response - target lesions) and/or, enlargement of non-target lesions.
Time Frame: up to 4 years
Reporting Status: Not Posted

5. Secondary Outcome: Change in CD45 Cells
Description: Within-patient mean change in percent of total number of CD45 cells present in tumor tissue and peritoneal fluid from treatment Cycle 1 Day 1.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 6.8 (44.6)

6. Secondary Outcome: Change in CD45 Cells
Description: as for outcome 5
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 21.5 (13.8)

7. Secondary Outcome: Change in CD45 Cells
Description: as for outcome 5
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 28.4 (19.3)

8. Secondary Outcome: Percent of CD45 Cells
Description: Mean percent of total CD45 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 7
percentage of cells | 57.9 (28.9)

9. Secondary Outcome: Percent of CD45 Cells
Description: Mean percent of total CD45 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 76 (32)

10. Secondary Outcome: Percent of CD45 Cells
Description: Mean percent of total CD45 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 91.3 (6.5)

11. Secondary Outcome: Percent of CD45 Cells
Description: Mean percent of total CD45 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 90.5 (8.5)

12. Secondary Outcome: Change in CD3 Cells
Description: Within-patient mean change in percent of total number of CD3 cells present in tumor tissue and peritoneal fluid from treatment Cycle 1 Day 1.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | -14.4 (13.8)

13. Secondary Outcome: Change in CD3 Cells
Description: as for outcome 12
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 22.5 (15.6)

14. Secondary Outcome: Change in CD3 Cells
Description: as for outcome 12
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | -7.8 (19.8)

15. Secondary Outcome: Percent of CD3 Cells
Description: Mean percent of total CD3 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 7
percentage of cells | 17.9 (13.9)

16. Secondary Outcome: Percent of CD3 Cells
Description: Mean percent of total CD3 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 4.5 (2.5)

17. Secondary Outcome: Percent of CD3 Cells
Description: Mean percent of total CD3 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 50.8 (20.3)

18. Secondary Outcome: Percent of CD3 Cells
Description: Mean percent of total CD3 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 10.5 (6.3)

19. Secondary Outcome: Change in CD4 Cells
Description: Within-patient mean change in percent of total number of CD4 cells present in tumor tissue and peritoneal fluid from treatment Cycle 1 Day 1.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | -5.9 (10.8)

20. Secondary Outcome: Change in CD4 Cells
Description: as for outcome 19
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 2 (28.6)

21. Secondary Outcome: Change in CD4 Cells
Description: as for outcome 19
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | -6.2 (12.4)

22. Secondary Outcome: Percent of CD4 Cells
Description: Mean percent of total CD4 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 7
percentage of cells | 6.9 (10.7)

23. Secondary Outcome: Percent of CD4 Cells
Description: Mean percent of total CD4 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 1.4 (1.2)

24. Secondary Outcome: Percent of CD4 Cells
Description: Mean percent of total CD4 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 14.5 (16.4)

25. Secondary Outcome: Percent of CD4 Cells
Description: Mean percent of total CD4 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 2.4 (1.7)

26. Secondary Outcome: Change in CD8 Cells
Description: Within-patient mean change in percent of total number of CD8 cells present in tumor tissue and peritoneal fluid from treatment Cycle 1 Day 1.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | -4.5 (6.3)

27. Secondary Outcome: Change in CD8 Cells
Description: as for outcome 26
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | -0.4 (2.1)

28. Secondary Outcome: Change in CD8 Cells
Description: as for outcome 26
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | -5 (7.8)

29. Secondary Outcome: Percent of CD8 Cells
Description: Mean percent of total CD8 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 7
percentage of cells | 5.7 (5.9)

30. Secondary Outcome: Percent of CD8 Cells
Description: Mean percent of total CD4 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 1.2 (0.8)

31. Secondary Outcome: Percent of CD8 Cells
Description: Mean percent of total CD8 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 11.9 (8.6)

32. Secondary Outcome: Percent of CD8 Cells
Description: Mean percent of total CD8 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 2.3 (2.3)

33. Secondary Outcome: Change in CD14 Cells
Description: Within-patient mean change in percent of total number of CD14 cells present in tumor tissue and peritoneal fluid from treatment Cycle 1 Day 1.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Median (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 36.8 (39.9)

34. Secondary Outcome: Change in CD14 Cells
Description: as for outcome 33
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Median (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | -20.6 (26.3)

35. Secondary Outcome: Change in CD14 Cells
Description: as for outcome 33
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Median (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 16.4 (36.1)

36. Secondary Outcome: Percent of CD14 Cells
Description: Mean percent of total CD14 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 7
percentage of cells | 15.5 (18.8)

37. Secondary Outcome: Percent of CD14 Cells
Description: Mean percent of total CD14 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 60.9 (29.1)

38. Secondary Outcome: Percent of CD14 Cells
Description: Mean percent of total CD14 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 6.7 (1.8)

39. Secondary Outcome: Percent of CD14 Cells
Description: Mean percent of total CD14 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 55.7 (29)

40. Secondary Outcome: Change in CD19 Cells
Description: Within-patient mean change in percent of total number of CD19 cells present in tumor tissue and peritoneal fluid from treatment Cycle 1 Day 1.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | -0.7 (1.4)

41. Secondary Outcome: Change in CD19 Cells
Description: as for outcome 40
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | -0.5 (0.1)

42. Secondary Outcome: Change in CD19 Cells
Description: as for outcome 40
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | -1.1 (1.7)

43. Secondary Outcome: Percent of CD19 Cells
Description: Mean percent of total CD19 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 7
percentage of cells | 1.1 (1.5)

44. Secondary Outcome: Percent of CD19 Cells
Description: Mean percent of total CD19 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 0.6 (0.4)

45. Secondary Outcome: Percent of CD19 Cells
Description: Mean percent of total CD19 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 1.5 (1.9)

46. Secondary Outcome: Percent of CD19 Cells
Description: Mean percent of total CD19 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 0.4 (0.2)

47. Secondary Outcome: Change in CD56 Cells
Description: Within-patient mean change in percent of total number of CD56 cells present in tumor tissue and peritoneal fluid from treatment Cycle 1 Day 1.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | -2 (3)

48. Secondary Outcome: Change in CD56 Cells
Description: as for outcome 47
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | -1.4 (1.8)

49. Secondary Outcome: Change in CD56 Cells
Description: as for outcome 47
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | -1.9 (3.1)

50. Secondary Outcome: Percent of CD56 Cells
Description: Mean percent of total CD56 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 7
percentage of cells | 2.9 (3.4)

51. Secondary Outcome: Percent of CD56 Cells
Description: Mean percent of total CD56 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 1 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 14
percentage of cells | 1.1 (0.9)

52. Secondary Outcome: Percent of CD56 Cells
Description: Mean percent of total CD56 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 1
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 4
percentage of cells | 4.2 (3)

53. Secondary Outcome: Percent of CD56 Cells
Description: Mean percent of total CD56 cells present in tumor tissue and peritoneal fluid from treatment.
Time Frame: At treatment Cycle 4 Day 3
Population: Treated patients who provided analyzable samples.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
Number analyzed (Participants) | 12
percentage of cells | 1.3 (0.9)

54. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2027-01

55. Other Pre Specified Outcome: NK Cells
Time Frame: at baseline (pre-treatment) and at 12 weeks (after the start of treatment)
Reporting Status: Not Posted

56. Other Pre Specified Outcome: Grandzyme B
Time Frame: at baseline (pre-treatment) and at 12 weeks (after the start of treatment)
Reporting Status: Not Posted

57. Other Pre Specified Outcome: CD4 Tbet
Time Frame: at baseline (pre-treatment) and at 12 weeks (after the start of treatment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events data collected for 5 years, 1 month All-Cause Mortality data provided to date; data still being collected.
Arm/Group | Cisplatin + Rintatolimod + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 12/24
Serious Adverse Events (participants affected / at risk) | 9/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Rintatolimod + Pembrolizumab (N=24)
Vomiting (GASTROINTESTINAL DISORDERS) | 1
Small intestinal perforation (GASTROINTESTINAL DISORDERS) | 1
Small intestinal obstruction (GASTROINTESTINAL DISORDERS) | 1
Obstruction gastric (GASTROINTESTINAL DISORDERS) | 1
Nausea (GASTROINTESTINAL DISORDERS) | 1
Abdominal pain (GASTROINTESTINAL DISORDERS) | 2
Fever (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2
Fatigue (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1
Sepsis (INFECTIONS AND INFESTATIONS) | 1
Device related infection (INFECTIONS AND INFESTATIONS) | 1
Hyponatremia (METABOLISM AND NUTRITION DISORDERS) | 1
Hypokalemia (METABOLISM AND NUTRITION DISORDERS) | 1
Hyperglycemia (METABOLISM AND NUTRITION DISORDERS) | 2
Dehydration (METABOLISM AND NUTRITION DISORDERS) | 1
Erythema multiforme (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Failure to thrive (SOCIAL CIRCUMSTANCES) | 1
Hypotension (VASCULAR DISORDERS) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Rintatolimod + Pembrolizumab (N=24)
Febrile neutropenia (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 2
Anemia (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 19
Sinus tachycardia (CARDIAC DISORDERS) | 6
Sinus bradycardia (CARDIAC DISORDERS) | 2
Palpitations (CARDIAC DISORDERS) | 1
Vertigo (EAR AND LABYRINTH DISORDERS) | 1
Tinnitus (EAR AND LABYRINTH DISORDERS) | 3
Adrenal insufficiency (ENDOCRINE DISORDERS) | 1
Watering eyes (EYE DISORDERS) | 2
Eye pain (EYE DISORDERS) | 1
Blurred vision (EYE DISORDERS) | 1
Vomiting (GASTROINTESTINAL DISORDERS) | 8
Small intestinal perforation (GASTROINTESTINAL DISORDERS) | 1
Small intestinal obstruction (GASTROINTESTINAL DISORDERS) | 1
Oral dysesthesia (GASTROINTESTINAL DISORDERS) | 1
Obstruction gastric (GASTROINTESTINAL DISORDERS) | 1
Nausea (GASTROINTESTINAL DISORDERS) | 20
Gastrointestinal pain (GASTROINTESTINAL DISORDERS) | 2
Bloody stools (GASTROINTESTINAL DISORDERS) | 1
Gastroesophageal reflux disease (GASTROINTESTINAL DISORDERS) | 1
Dysphagia (GASTROINTESTINAL DISORDERS) | 1
Dyspepsia (GASTROINTESTINAL DISORDERS) | 1
Dry mouth (GASTROINTESTINAL DISORDERS) | 3
Diarrhea (GASTROINTESTINAL DISORDERS) | 12
Constipation (GASTROINTESTINAL DISORDERS) | 5
Bloating (GASTROINTESTINAL DISORDERS) | 12
Ascites (GASTROINTESTINAL DISORDERS) | 1
Abdominal pain (GASTROINTESTINAL DISORDERS) | 16
Abdominal distension (GASTROINTESTINAL DISORDERS) | 3
Pain (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 6
Infusion site extravasation (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1
Flu like symptoms (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1
Fever (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2
Fatigue (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 24
Edema limbs (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1
Chills (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 4
Allergic reaction (IMMUNE SYSTEM DISORDERS) | 1
Vaginal infection (INFECTIONS AND INFESTATIONS) | 1
Urinary tract infection (INFECTIONS AND INFESTATIONS) | 4
Upper respiratory infection (INFECTIONS AND INFESTATIONS) | 2
Skin infection (INFECTIONS AND INFESTATIONS) | 1
Sepsis (INFECTIONS AND INFESTATIONS) | 1
Device related infection (INFECTIONS AND INFESTATIONS) | 1
Bacteremia (INFECTIONS AND INFESTATIONS) | 1
Abdominal infection (INFECTIONS AND INFESTATIONS) | 1
Infusion related reaction (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1
Fall (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 2
Bruising (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1
White blood cell decreased (INVESTIGATIONS) | 7
Weight loss (INVESTIGATIONS) | 2
Platelet count decreased (INVESTIGATIONS) | 3
Neutrophil count decreased (INVESTIGATIONS) | 10
Lymphocyte count decreased (INVESTIGATIONS) | 8
increased BUN (INVESTIGATIONS) | 1
Creatinine increased (INVESTIGATIONS) | 5
Blood lactate dehydrogenase increased (INVESTIGATIONS) | 7
Aspartate aminotransferase increased (INVESTIGATIONS) | 4
Alkaline phosphatase increased (INVESTIGATIONS) | 3
Hypophosphatemia (METABOLISM AND NUTRITION DISORDERS) | 5
Hyponatremia (METABOLISM AND NUTRITION DISORDERS) | 13
Hypomagnesemia (METABOLISM AND NUTRITION DISORDERS) | 21
Hypokalemia (METABOLISM AND NUTRITION DISORDERS) | 5
Hypoglycemia (METABOLISM AND NUTRITION DISORDERS) | 2
Hypocalcemia (METABOLISM AND NUTRITION DISORDERS) | 2
Hypoalbuminemia (METABOLISM AND NUTRITION DISORDERS) | 3
Hyperuricemia (METABOLISM AND NUTRITION DISORDERS) | 1
Hyperglycemia (METABOLISM AND NUTRITION DISORDERS) | 6
Hypercalcemia (METABOLISM AND NUTRITION DISORDERS) | 1
Dehydration (METABOLISM AND NUTRITION DISORDERS) | 3
Anorexia (METABOLISM AND NUTRITION DISORDERS) | 11
Myalgia (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1
Generalized muscle weakness (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3
Back pain (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 5
Arthralgia (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3
Tremor (NERVOUS SYSTEM DISORDERS) | 4
Syncope (NERVOUS SYSTEM DISORDERS) | 1
Peripheral sensory neuropathy (NERVOUS SYSTEM DISORDERS) | 3
Peripheral motor neuropathy (NERVOUS SYSTEM DISORDERS) | 1
Lethargy (NERVOUS SYSTEM DISORDERS) | 2
Headache (NERVOUS SYSTEM DISORDERS) | 7
Dysgeusia (NERVOUS SYSTEM DISORDERS) | 1
Dizziness (NERVOUS SYSTEM DISORDERS) | 3
Akathisia (NERVOUS SYSTEM DISORDERS) | 1
Claustrophobic (PSYCHIATRIC DISORDERS) | 1
Insomnia (PSYCHIATRIC DISORDERS) | 2
Confusion (PSYCHIATRIC DISORDERS) | 1
Anxiety (PSYCHIATRIC DISORDERS) | 1
Urinary incontinence (RENAL AND URINARY DISORDERS) | 1
Urinary frequency (RENAL AND URINARY DISORDERS) | 1
Proteinuria (RENAL AND URINARY DISORDERS) | 2
Hematuria (RENAL AND URINARY DISORDERS) | 3
Chronic kidney disease (RENAL AND URINARY DISORDERS) | 3
Pelvic pain (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1
Rhinorrhea (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1
Postnasal drip (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2
Nasal congestion (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 7
Hiccups (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1
Dyspnea (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2
Cough (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 3
Skin redness/ irritation (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
RUQ Redness/ Irritation (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Dermatologic Toxicity (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Cellulitus (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Rash maculo-papular (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 4
Rash acneiform (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Pruritus (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2
Hyperhidrosis (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Erythema multiforme (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Bullous dermatitis (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2
Alopecia (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1
Failure to thrive (SOCIAL CIRCUMSTANCES) | 1
Thromboembolic event (VASCULAR DISORDERS) | 1
Hypotension (VASCULAR DISORDERS) | 5
Hypertension (VASCULAR DISORDERS) | 15
Hematoma (VASCULAR DISORDERS) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03734692/Prot_SAP_000.pdf